CLINICAL TRIAL: NCT06689046
Title: Nausea and Vomiting Following Esophagogastroduodenoscopy: Prevalence and Predictive Factors
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Gülencan Yumuşak Ergin, Consultant anesthesiologist, Aksaray University Training and Research Hospital
Other Study IDs: 2023/23-37
Record Dates: First submitted 2024-11-10; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Nausea and Vomiting; Esophagogastroduodenoscopy
Keywords: postoperative nausea and vomiting; esophagogastroduodenoscopy
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endoscopic procedures are widely implemented to diagnose both malignant and benign diseases. Nausea and vomiting is a common complication after anesthesia. Yet, nausea and vomiting after endoscopic procedures are not dully established.

The primary aim of the study is to assess the incidence of postoperative nausea and vomiting in patients who underwent esophagogastroduodenoscopy. The secondary aim is to identify possible risk factors, both related to the patients and the procedure itself.

DETAILED DESCRIPTION:
Nausea, vomiting, and retching are common issues that can complicate recovery after anesthesia. Many patients regard these experiences as unpleasant and reduce the quality of life and quality of recovery of patients. It has been suggested to increase healthcare costs due to prolonged length of stay, readmissions, and possibly life-threatening adverse effects such as pulmonary aspiration and aspiration pneumonia [1-3]. These unwanted consequences make postoperative nausea and vomiting (PONV) one of the most important issues for anesthesiologists.

PONV typically resolves on its own or can be effectively treated without lasting effects. Many studies have been carried out to identify prevalence and risk factors [4, 5]. The occurrence of PONV can vary depending on surgery, anesthesia, and patient characteristics. Generally, about 30% of patients undergoing surgery experience PONV, but this rate can rise to as high as 80% in high-risk patients [6].

Numerous studies are focused on evaluating various measures aimed at reducing the prevalence, severity, and duration of nausea and vomiting throughout the perioperative period [7]. Apfel score is a simple, widely accepted tool to asses patients' PONV risk which consists of four independent risk factors such as non-smoker, female gender, history of PONV, history of motion sickness, and opioid usage in the postoperative period [8]. Koivuranta risk score, which is similar to the Apfel score, also includes age and duration of surgery [9]. Procedure-related risk factors are suggested to play a role in PONV. PONV is more common following laparoscopic, bariatric, and gynecological surgeries and cholecystectomies. Longer surgery duration, and using volatile agents and opioids are also related to PONV [10].

Nausea and vomiting can occur after gastrointestinal endoscopic procedures due to the excessive stretching of the stomach and intestinal loops [11]. Wu et al. suggested that the rates of nausea and vomiting after endoscopic procedures were 4.1% and 2.9%, respectively. Wu and colleagues also observed that the female gender is an independent risk factor for developing PONV [12]. Hormati et al. established that 1.42% of patients reported experiencing nausea and vomiting following various gastrointestinal endoscopic procedures [13]. They noted that postoperative nausea and vomiting (PONV) was the second most common complication, following hemodynamic instability. Although endoscopic procedures are frequently performed around the globe, and also PONV is a common and possibly dangerous complication, the frequency and risk factors of developing PONV after endoscopic procedures have not been fully determined. The primary aim of the study is to assess the incidence of postoperative nausea and vomiting in patients who underwent esophagogastroduodenoscopy. An additional goal is to identify possible risk factors, both related to the patients and the procedure itself.

ELIGIBILITY:
Inclusion Criteria:

* having an endoscopic procedure with sedation

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had undergone an endoscopic procedure with sedation
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of Nausea and Vomiting following Esophagogastroduodenoscopy | post procedure day 1
  Prevalence of Nausea and Vomiting following Esophagogastroduodenoscopy

SECONDARY OUTCOMES:
Risk Factors of Nausea and Vomiting following Esophagogastroduodenoscopy | post procedure day 1
  Risk Factors of Nausea and Vomiting following Esophagogastroduodenoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Aksaray University, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parra-Sanchez I, Abdallah R, You J, Fu AZ, Grady M, Cummings K 3rd, Apfel C, Sessler DI. A time-motion economic analysis of postoperative nausea and vomiting in ambulatory surgery. Can J Anaesth. 2012 Apr;59(4):366-75. doi: 10.1007/s12630-011-9660-x. Epub 2012 Jan 6. PMID 22223185